CLINICAL TRIAL: NCT05846009
Title: A Phase I, First-in-human, Two-part, Randomized, Placebo-controlled, Double-blind, Single and Repeated Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous Doses of SAR442501 in Healthy Adult Subjects
Brief Title: A First-in-human Single and Repeated Dose Escalation Study of SAR442501 in Healthy Adults Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TDU16639/TDR16640
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Osteochondrodysplasia
MeSH Terms: conditions — Osteochondrodysplasias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR442501 (Experimental)
  Interventions: Drug: SAR442501
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR442501 — Subcutaneous injection
  Arms: SAR442501
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of the first-in-human (FIH) study is to obtain safety, tolerability, and pharmacokinetic information on SAR442501 in a healthy adult volunteer population using an integrated single ascending dose (SAD)-multiple ascending dose (MAD) parallel cohort study design.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, between 18 and 45 years of age, inclusive.
* Body weight between 50.0 and 85.0 kg, inclusive, body mass index between 18.0 and 32.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* Any history or presence of clinically relevant medical status as per the protocol.
* Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events/treatment-emergent adverse events/adverse events of special interest | Baseline up to end of study (EOS) (Day 89)

SECONDARY OUTCOMES:
Assessment of PK parameter: Maximum observed concentration (Cmax) | Baseline up to EOS (Day 89)
Assessment of PK parameter: First time to reach Cmax (tmax) | Baseline up to EOS (Day 89)
Assessment of PK parameter: Partial area under the serum concentration time curve (AUC) | Baseline up to EOS (Day 89)
Immunogenicity: evaluate the presence of anti-SAR442501 antibodies | Baseline up to EOS (Day 89)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TDU16639/TDR16640 Plain language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25464&tenant=MT_SNY_9011